CLINICAL TRIAL: NCT03102645
Title: Effect of Single Dose Imipramine on the Urethral and Anal Sphincter in Healthy Women Measured With Urethral Pressure Reflectometry (UPR) and Anal Acoustic Reflectometry (AAR)
Brief Title: Does Single Dose Imipramine Affect the Opening Pressure of the Urethral and Anal Sphincter?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonatan Kornholt (Other)
Responsible Party: Sponsor-Investigator, Jonatan Kornholt, Resident doctor in the Department of Clinical Pharmacology, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: TCA-UPR-0001
Record Dates: First submitted 2017-03-20; First posted 2017-04-06 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence, Stress; Fecal Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Fecal Incontinence | interventions — Imipramine

STUDY DESIGN:
Intervention Model Description: 16 healthy female subjects. Double-blinded, crossover study on two days with 1 week washout. Either placebo or imipramine 50 mg single dose before and after measurement of UOP and AOP.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Packaging, randomization and masking of investigational drugs (imipramine and placebo) by Region Hovedstadens Apothecary before delivery to investigator. Sealed envelope with participant ID and drug data will be opened after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imipramine first (Experimental): A: Imipramine Hydrochloride 25 MG x2 B: Placebo Oral Tablet x2
  Interventions: Drug: Placebo Oral Tablet; Drug: Imipramine Hydrochloride 25 MG
- Placebo first (Experimental): A: Placebo Oral Tablet x2 B: Imipramine Hydrochloride 25 MG x2
  Interventions: Drug: Placebo Oral Tablet; Drug: Imipramine Hydrochloride 25 MG

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo film coated tablet: Lactose monohydrate, potato starch, gelatine, magnesium stearate, talc
Drug: Imipramine Hydrochloride 25 MG — Two Imipramin DAK film coated tablets 25 mg each, single dose
  Other Names: Imipramin DAK

SUMMARY:
A double-blinded, randomized, crossover study in healthy females with placebo and single dose imipramine 50 mg.

Primary objective: Does imipramine increase the tone of the external urethral sphincter? Urethral Opening Pressure (UOP) is measured with Urethral Pressure Reflectometry (UPR). UOP increases correlate with effect in treating stress urinary incontinence. Can imipramine treat stress urinary incontinence? Secondary objective: Does imipramine increase the tone of the anal sphincter? The opening pressure is measured with Anal Acoustic Reflectometry (AAR). The investigators also wish to establish the within-subject standard deviation for AAR to enable power calculations in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form.
* Healthy.
* Female.
* Non-smoker.
* Age 18 to 55, both inclusive.
* Normal weight: BMI 19.5 to 30.0 kg/m2. Weight minimum 50 kg.
* No breastfeeding.
* No pregnancy during the study.
* No other clinical trials during the study.

Exclusion Criteria:

* Known allergy to imipramine or any of the other known constituents.
* Medical history with significant cardiovascular, gastrointestinal, endocrinologic, hematologic, immunologic, metabolic, genitourologic, dermatologic, psychiatric, neurologic or dermatologic disease, lung disease, kidney disease, malignant disease or other significant diseases as assessed by the investigator.
* Medical history of urinary incontinence.
* Infectious disease 1 week prior to study day 1 or study day 2.
* Clinically significant findings during the physical examination.
* Pregnancy.
* Heart rate < 40 or > 100 beats per minute. Mean systolic blood pressure > 140 mmHg or mean diastolic blood pressure > 90 mmHg (mean of the measures on the screening day).
* Prescription, over the counter or herbal medication two weeks prior to study day 1 or study day 2. Excluding paracetamol and excluding oral contraceptives.
* Smoking 3 months prior to study day 1 or study day 2.
* Alcohol abuse, meaning > 14 units (12 g alcohol) per week within three weeks prior to study day 1 or study day 2.
* Drug abuse 3 months prior to study day 1 or study day 2.
* Any condition as assessed by the investigator.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Kornholt, MD, Principal Investigator — Klinisk farmakologisk afdeling, Bispebjerg Hospital
Locations (1):
- Zelo Phase I Unit, Dept. of Clinical Pharmacology, Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were included from 16 May 2017 to 31 May 2017 and the study days was conducted from 17 May 2017 to 16 June 2017 and the last followup call to detect adverse effects was 21 June 2017.
Pre-assignment Details: Randomization determining order of arms after enrollment. At least 1 week wash out between study days. Followup 5 days after last study day to collect adverse events.
Period: Overall Study
Arm/Group | Imipramine First | Placebo First
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imipramine First | Placebo First | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Urethral Opening Pressure (UOP)
Description: Mean change in UOP (baseline and 1 hour after drug administration). Measured with Urethral Pressure Reflectometry (UPR).
Time Frame: Immediately before drug/placebo administration (baseline) and 1 hour after drug/placebo administration on both study days.
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Imipramine: Imipramine Hydrochloride 25 MG: Two Imipramin DAK film coated tablets 25 mg each, single dose.
- Placebo: Placebo Oral Tablet: Placebo film coated tablet: Lactose monohydrate, potato starch, gelatine, magnesium stearate, talc
Arm/Group | Imipramine | Placebo
Number analyzed (Participants) | 16 | 16
cmH2O | 2.90411 (13.24729) | -3.623431 (8.279883)
Statistical Analysis 1: Comparison: Imipramine vs Placebo; CROS test; Test type: Superiority; p = 0.07, t-test, 2 sided; CROS. DF=14; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [-0.5 to 13.5]

2. Secondary Outcome: Anal Opening Pressure (AOP)
Description: Mean change in AOP (baseline and 1 hour after drug administration). Measured with Anal Acoustic Reflectometry (AAR).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Imipramine | Placebo
Number analyzed (Participants) | 16 | 16
cmH2O | 12.11873 (15.79818) | -2.989054 (16.40355)
Statistical Analysis 1: Comparison: Imipramine vs Placebo; CROS test; Test type: Superiority; p = 0.03, t-test, 2 sided; CROS test; Mean Difference (Final Values) = 15.2, 95% CI 2-sided [2.0 to 28.2]

ADVERSE EVENTS:
Time Frame: From study day 1 to 5 days after 2nd study day.
Groups:
- Imipramine: Imipramine Hydrochloride 25 MG x2: Two Imipramin DAK film coated tablets 25 mg each, single dose
- Placebo: Placebo Oral Tablet x2: Two placebo film coated tablets containing lactose monohydrate, potato starch, gelatine, magnesium stearate, and talc
Arm/Group | Imipramine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imipramine (N=16) | Placebo (N=16)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Tired (General disorders) | 5 (5) | 0 (0)
Dizzy (Nervous system disorders) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03102645/Prot_SAP_000.pdf